CLINICAL TRIAL: NCT05910099
Title: Investigating Medical Research Trends in Rectal Cancer Clinical Study: Analyzing Factors Impacting Patient Involvement
Brief Title: Taking a Look at Patient Experiences In Rectal Cancer Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85996123
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this research study is to explore the barriers encountered by specific demographic groups of rectal cancer patients during the engagement in clinical trials, which historically lack diverse representation.

By carefully analyzing data from various demographic perspectives, this study aims to uncover patterns that impact the experiences of future rectal cancer patients. Active involvement in this crucial research is of utmost importance, as it can offer unique insights to enhance the participation and completion rates of rectal cancer patients in clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of rectal cancer
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* No prior treatment for rectal cancer

Exclusion Criteria:

* Pregnant or lactating woman
* Inability to provide written informed consent
* Enrolled in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer who are actively participating in a clinical research, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of rectal cancer patients who decide to participate in a clinical study | 3 months
Rate of patients who remain in a rectal cancer clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvarez Sarrado E, Giner Segura F, Batista Domenech A, Garcia-Granero Garcia-Fuster A, Frasson M, Rudenko P, Flor Lorente B, Garcia-Granero Ximenez E. Rectal cancer at the peritoneal reflection. Preoperative MRI accuracy and histophatologic correlation. Prospective study. Cir Esp (Engl Ed). 2022 Aug;100(8):488-495. doi: 10.1016/j.cireng.2022.05.019. Epub 2022 May 18. PMID 35597413
- [Background] Bregendahl S, Bondeven P, Gronborg TK, Brown G, Laurberg S, Pedersen BG. Training of radiology specialists in local staging of primary rectal cancer on MRI: a prospective intervention study exploring the impact of various educational elements on the interpretive performance. BMJ Open Qual. 2022 Aug;11(3):e001716. doi: 10.1136/bmjoq-2021-001716. PMID 35944932
- [Background] Qaderi SM, Dickman PW, de Wilt JHW, Verhoeven RHA. Conditional Survival and Cure of Patients With Colon or Rectal Cancer: A Population-Based Study. J Natl Compr Canc Netw. 2020 Sep;18(9):1230-1237. doi: 10.6004/jnccn.2020.7568. PMID 32886900

DOCUMENTS (1):
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT05910099/ICF_000.pdf